CLINICAL TRIAL: NCT06122077
Title: The PROACT LUNG Study: A Prospective, Observational,Clinical Validation Study of the Freenome Multiomics Blood Test for Lung Cancer Screening (FRNM-007)
Brief Title: Clinical Validation of Freenome Multiomics Blood Test for Lung Cancer Screening
Acronym: PROACT-LUNG
Status: Recruiting | Type: Observational
Sponsor: Freenome Holdings Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FRNM-007
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer Diagnosis
Keywords: Artificial Intelligence; Liquid Biopsy; Blood Test Cancer; Cancer Diagnostic; Genomics; Genomics Test; Multiomics; Cancer Screening; Cancer Early Detection Test; LDCT Screening; Lung Cancer Screening; Lung Cancer; Freenome Test; Machine Learning; Acute respiratory distress syndrome (ARDS); Chronic obstructive pulmonary disease (COPD); Chronic bronchitis; Emphysema; Lung nodules
MeSH Terms: conditions — Lung Neoplasms; Respiratory Distress Syndrome; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be de-identified and used to validate the performance characteristics of the Freenome Multiomics Blood Test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Diagnostic Test: blood draw — Subjects who provide informed consent and meet the eligibility criteria will have 50 ml of blood collected and sent to Freenome or Freenome's designee for processing, testing, and storage, and will then complete a standard-of-care screening LDCT.

SUMMARY:
The PROACT LUNG study is a prospective multi-center observational study to validate a blood-based test for the early detection of lung cancer by collecting blood samples from high-risk participants who will undergo a routine, standard-of-care screening Low-Dose Computed Tomography (LDCT).

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study to evaluate the performance of the Freenome Multiomics Blood Test in screening eligible participants for lung cancer.

Enrollment will be open to all eligible participants for screening chest CT scan as part of the Standard of Care (SOC) for lung cancer. Subjects who meet the eligibility criteria for this study and provide informed consent will be enrolled and blood sample collection must be completed within 30 days of signing the informed consent. Optimally, the screening chest CT will be completed on the same day of the study blood collection, however up to 45 days will be allowed after study blood collection to obtain a screening chest CT.

The study will also collect demographic data and relevant clinical data, such as medical history, lifestyle, occupational and environmental exposure(s), family history, and clinical laboratory data. All reports and clinical notes regarding the diagnostic tests and procedures related to lung cancer diagnosis or lung lesion assessment, such as histopathology and bronchoscopy reports, and diagnostic/follow-up images and imaging reports will be collected as part of follow up to the screening chest CT scan.

All enrolled subjects will be followed prospectively from the date of the baseline screening chest CT until a minimum of 24 months, or until a premature study endpoint inclusive of withdrawal of consent or death.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years or older within 30 days of enrollment
2. Current or former smokers with a cumulative smoking history of ≥ 20 pack-year
3. Able to comprehend and willing to sign and date the informed consent and HIPAA authorization documents

Exclusion Criteria:

1. Any active therapy for cancer, including but not limited to surgery, chemotherapy, biologic therapy, immunotherapy, and/or radiation therapy at the time of enrollment
2. History of any malignancy within prior 5 years of enrollment (except for non- melanoma skin cancer)
3. History of organ, tissue, and bone marrow transplantation
4. Screened for lung cancer or having chest CT scan 12 months before enrollment
5. Having signs and symptoms of lung cancer such as hemoptysis, superior vena cava syndrome, Cushing syndrome, and Pancoast syndrome
6. Received a blood transfusion in the 30 days preceding enrollment
7. Known to be pregnant
8. Participated or currently participating in another Freenome-sponsored clinical study
9. Participated or currently participating in a clinical research study in which an experimental medication has been administered during the 60 days preceding enrollment
10. Any condition that in the opinion of the Investigator should not be enrolled in the study

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex assigned at birth
Study Population: The study aims to enroll a representative sample of the population across the United States including adults aged 50 years and older who have at least a 20-pack-year smoking history and who have met the eligibility criteria defined in this protocol.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity in detecting lung cancer | 12-Months
  Clinical performance of the Freenome Blood Test, including sensitivity and specificity, in detecting lung cancer in subjects with positive and negative lung cancer outcomes during a 12-month follow-up period

SECONDARY OUTCOMES:
Sensitivity and specificity in detecting lung cancer | 24-Months
  Clinical performance of the Freenome Blood Test, including sensitivity and specificity, in detecting lung cancer in subjects with positive and negative lung cancer outcomes during a 24-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Sumner, Study Director — Freenome Holdings Inc.
Locations (36):
- United States (36):
  - Science 37, Los Angeles, California
  - Stamford Hospital, Stamford, Connecticut
  - Hillcrest Medical Research, DeLand, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - I.H.S Health, LLC, Kissimmee, Florida
  - United Medical Research, Port Orange, Florida
  - Charter Research, The Villages, Florida
  - Charter Research, Winter Park, Florida
  - SpeciCare, Inc, Gainesville, Georgia
  - University of Chicago, Chicago, Illinois
  - Walgreens, Deerfield, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Aton Health, Leawood, Kansas
  - Ascension Via Christi Wichita, Wichita, Kansas
  - Ascension St. Agnes Hospital, Baltimore, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Renown Regional Medical Center, Reno, Nevada
  - Inspira Medical Center, Mullica Hill, New Jersey
  - Our Lady of Lourdes Hospital, Binghamton, New York
  - Wakemed, Raleigh, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Clinical Research Associates of Central PA, DuBois, Pennsylvania
  - US Digestive Health at Lancaster, Lancaster, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Guthrie Medical Group, Sayre, Pennsylvania
  - US Digestive Health at Wyomissing, Wyomissing, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - McLeod Health, Florence, South Carolina
  - Circle Clinical Research, Pierre, South Dakota
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Horizon Clinical Research Group, Houston, Texas
  - CHRISTUS Trinity Mother Frances Health System, Tyler, Texas
  - Ascension Columbia St. Mary's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No